CLINICAL TRIAL: NCT01363817
Title: Phase 1 Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of BMS-906024 in Subjects With Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma
Brief Title: Study to Evaluate the Safety and Tolerability of Weekly Intravenous (IV) Doses of BMS-906024 in Subjects With Acute T-cell Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA216-002; 2010-022727-29 (EudraCT Number)
Record Dates: First submitted 2011-04-22; First posted 2011-06-02 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Lymphoblastic Leukemia, Acute T-cell; Precursor T-Cell Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — BMS-906024; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation Phase: BMS-906024 (Experimental): BMS-906024 escalating doses starting at 0.3 mg solution for intravenous (IV) administration once weekly continuously until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-906024
- Expansion Phase: BMS-906024 + Dexamethasone (Experimental): BMS-906024 maximum tolerated dose (To be determined) solution for IV administration once weekly and Dexamethasone 20mg/day tablet by mouth (Oral) for 3-4 days every week for 3-4 weeks per cycle continuously until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-906024; Drug: Dexamethasone

INTERVENTIONS:
Drug: BMS-906024
  Other Names: Notch inhibitor
Drug: Dexamethasone
  Other Names: Baycadron
  Arms: Expansion Phase: BMS-906024 + Dexamethasone

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of BMS-906024, either alone or in combination with Dexamethasone in subjects with T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma who no longer respond to or have relapsed from standard therapies

DETAILED DESCRIPTION:
Minimum Age: 10 years and older at selected sites

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma refractory to or relapsed from standard therapies
* Life expectancy of at least 2 months
* Performance status (PS) 0-1 (a measure of the ability to carry out activities of daily living); subjects with PS 2 are eligible if due to disease related symptoms
* Prior anti-cancer treatment permitted (with specific criteria)
* Adequate organ function

Exclusion Criteria:

* Infection
* Elevated triglycerides
* Gastro-intestinal disease with increased risk of diarrhea (e.g. inflammatory bowel disease)
* Unable to tolerate bone marrow biopsy
* Taking medications known to increase risk of Torsades De Pointes (an abnormal heart rhythm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09-28 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Weekly assessments until study discontinuation due to disease progression or unacceptable adverse events as well as an assessment 30 days after treatment discontinuation with an average time on study expected to be < 1 year.

SECONDARY OUTCOMES:
Disease assessments in bone marrow & by computed tomography (CT)/ magnetic resonance imaging (MRI) | Disease assessments at least every 8 weeks during treatment
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: maximum observed concentration (Cmax) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: minimum observed concentration (Cmin) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: area under the concentration-time curve (AUC) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: time to reach maximum observed concentration (Tmax) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: terminal phase elimination half-life (T-Half) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacokinetics of BMS-906024 and its metabolite BMS-911557: accumulation index (ratio of AUC at steady state to AUC after first dose) | Pharmacokinetics at multiple time points during the first 4 weeks of dosing
Pharmacodynamics (percent change from baseline in mRNA expression of Notch pathway-related genes in blood cells) | Pharmacodynamic sampling: in blood during the first 8 weeks of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Local Institution, Marseille
  - Local Institution, Paris
- Johann Wolfgang Goethe Universitaet, Frankfurt am Main, Germany

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx